CLINICAL TRIAL: NCT03410069
Title: Monitoring Tissue Perfusion in Critically Ill or High-risk Surgical Patients: a Pilot Clinical Study To Evaluate the aPplicability and the Safety of Urethral Perfusion Measurement With the IKORUS System
Brief Title: Monitoring Tissue Perfusion in Critically Ill or High-risk Surgical Patients
Acronym: STEP UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Perfusion Diagnostics (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A03466-47
Record Dates: First submitted 2018-01-12; First posted 2018-01-25 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: High-risk Surgical Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IKORUS UP (Experimental)
  Interventions: Device: IKORUS UP system

INTERVENTIONS:
Device: IKORUS UP system — Continuous assessment of the urethral microcirculation

SUMMARY:
Circulatory shock is defined as an imbalance between oxygen supply and/or impaired oxygen use to maintain organ function. With growing evidence of lack of correlation between macro- and micro-circulation, use of "Whole Body" markers such as blood pressure (BP) or Lactates are often insufficient to assess the severity of the oxygen debt and/or tissue hypoperfusion. Thus, an approach incorporating tissue-perfusion based endpoints would represent a significant step up to guide optimal resuscitation of critically-ill patients and to reduce complications in high-risk surgery.

Current monitoring techniques, that complement systemic hemodynamics by focusing on regional perfusion, still lack the required user-friendliness and/or clinical relevance to be routinely used at bedside. Therefore, assessment of the adequacy of tissue perfusion and oxygenation is suboptimal, and implementation of the above-mentioned approaches of resuscitation is still a challenge.

Urethral perfusion is likely to be early and significantly impaired during low-flow states and thus represents a good "candidate" as a surrogate site to assess the perfusion of visceral organs. Besides, urethral mucosa can be investigated in a less invasive and simpler manner than "deeper" organs. Nowadays, no practical methods or devices are available to monitor perfusion in the pelvic area. Thus, recent development of a new monitoring device of urethral perfusion could fill this need and enable enhanced management of patients in Intensive Care Units (ICU) and Operating Rooms (OR).

The device consists of a modified Foley catheter equipped with a photoplethysmographic sensor: the IKORUS UP probe.

The probe will be used by intensivists or anesthesiologists on high-risk surgical patients, i.e. patients with comorbidities undergoing major vascular, thoracic and/or abdominal surgery.

ELIGIBILITY:
Inclusion criteria:

1. 18 years of age or more,
2. Male or female,
3. High-Risk surgical patient,
4. Life expectancy expected to exceed 72 hours,
5. Willing to participate and signed informed consent,
6. Affiliation to the French social security system.

Non inclusion criteria:

1. Pregnant or lactating woman,
2. History of recent urological surgery (bladder surgery, prostate surgery…),
3. Known stricture or "impossible insertion" last hospitalization,
4. Traumatic injury to the lower urinary tract,
5. History of radiotherapy of pelvic or genital area,
6. Genital malformation (Hypospadias…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | 28 days
  Complications rate: Injury during insertion; Bleeding; Infection; Pain; Discomfort.

SECONDARY OUTCOMES:
Applicability of the procedure | 28 days
  Evaluation of applicability (compared to a standard Foley catheter): questionnaire for the nurse and/or the physician.
Signal acquisition | 28 days
  Duration of useable signal acquisition (duration of perfusion index computation)
Effect of the position of the sensor | 28 days
  Quality of signal according to sensor position (proximal/distal)
Quality of the signal | 28 days
  Assessment of signal Quality, including Signal-to-noise ratio
Evolution of mean arterial pressure | 28 days
  Measures of hemodynamic /metabolic parameters: mean arterial pressure (MAP)
Evolution of SpO2 | 28 days
  Measures of hemodynamic /metabolic parameters: SpO2
Evolution of SVO2 | 28 days
  Measures of hemodynamic /metabolic parameters: SVO2
Evolution of lactates dosages | 28 days
  Measures of hemodynamic /metabolic parameters: lactactes
Evolution of cardiac outputs | 28 days
  Measures of hemodynamic /metabolic parameters: cardiac output
Evolution of central venous pressure | 28 days
  Measures of hemodynamic /metabolic parameters: central venous pressure (CVP)
Evolution of catecholamine infusions levels | 28 days
  Measures of hemodynamic /metabolic parameters: catecholamine infusions levels
Rate of resuscitation events | 28 days
  Measures of hemodynamic or metabolic parameters: resuscitation events

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Allaouchiche, Prof, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - CHU Estaing, Clermont-Ferrand
  - Lyon Sud Hospital, Lyon
  - Hopital Nord Marseille, Marseille
  - Hospital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Depret F, Leone M, Duclos G, Futier E, Montagne M, Legrand M, Allaouchiche B. Monitoring tissue perfusion: a pilot clinical feasibility and safety study of a urethral photoplethysmography-derived perfusion device in high-risk patients. J Clin Monit Comput. 2020 Oct;34(5):961-969. doi: 10.1007/s10877-019-00414-9. Epub 2019 Nov 6. PMID 31691897